CLINICAL TRIAL: NCT03700814
Title: Comparison of Postoperative Infection and Graft Uptake Rate Using Single Dose of Intravenous Co-amoxiclav Versus no Antibiotic in Children Undergoing Myringoplasty
Brief Title: Does Antibiotics Use During Surgery Help to Decrease Wound Infection and Increase Success After Ear Surgery in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Prakash Khanal, ENT- Head and Neck Surgeon, Tribhuvan University, Nepal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121
Record Dates: First submitted 2018-09-29; First posted 2018-10-09 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Post Operative Wound Infection; Graft Uptake; Myringoplasty
MeSH Terms: conditions — Surgical Wound Infection | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotics group (Experimental): Patients in this group will receive single dose of intravenous co-amoxiclav (Dose: 25 mg/kg body weight) which will be injected 30 minutes prior to the incision during surgery.
  Interventions: Drug: Co-amoxiclav
- No antibiotics group (No Intervention): Patients belonging to this group will not receive any systemic antibiotic during intraoperative or post-operative period.

INTERVENTIONS:
Drug: Co-amoxiclav — Patients in this group will receive single dose of intravenous co-amoxiclav (Dose: 25 mg/kg body weight) which was injected 30 minutes prior to the incision during surgery.
  Arms: Antibiotics group

SUMMARY:
This study assess whether there is any role of antibiotics to decrease wound infection and increase the success of surgery

DETAILED DESCRIPTION:
Chronic Otitis Media is the disease of middle part of the ear. It presents with intermittent ear discharge and hearing loss of various severity. It is one of the commonest ear disease. This problem is treated with surgical procedure known as Myringoplasty. This surgical technique that involves repair of the tympanic membrane perforation. Myringoplasty is a clean type of surgery. Wound infection following this surgery is very low that is about less than 2 persons out of 100 people. So antibiotics is not necessary in this surgery. However antibiotics have been used unnecessarily. Unnecessary use of antibiotic increases financial burden to the patient and also leds to the development of drug resistant microorganisms.

The aims of this study is to evaluate the effectiveness and safety of antibiotics to decrease wound infection and increase the success of surgery. This will be a prospective, randomized, single-center, double-blinded, placebo controlled study. This study will be carried out over a period of 18 months from January 2014 to June 2015. The study will be carried out at Ganesh Man Singh Memorial Academy (GMSMA) of ENT-Head and Neck Studies, Tribhuvan University Teaching Hospital, Maharajgunj Medical Campus (MMC), Institute of Medicine (IOM), Kathmandu, Nepal.

Patient who are diagnosed to have chronic otitis media mucosal, inactive type who present in GMSMA of ENT- Head and Neck Studies outdoor clinic for surgery will be included for the study. Age of the patient included will be between six to 15 years of age. Both male and female patients can participate in this study. Patient who are having actively discharging ear cannot participate in the study. Similarly patients who are undergoing surgery for second times will not be qualified for study. Also patients who are allergic to co-amoxiclav will not be qualified for the study.

Total of sixty patients will participate in this study. The patients coming to our OPD will be first screened by the faculties Detail history, general physical examination, ENT - Head and Neck examination with Otoscopic examination and Tuning fork test will be done. Hearing assessment will be done. All patients will be admitted in ward day prior to surgery and pre-anaesthetic evaluation will be carried out by anaesthesiologist regarding their fitness for surgery under general anaesthesia.

Patients will be randomly divided in to two groups by lottery methods. However patient will not know about which group they belong. Patients in the first group will receive single dose of antibiotics which will be injected during surgery .Patients belonging to this group will not receive any antibiotics during surgery. All surgeries will be carried out under general anaesthesia by experienced faculty. Temporalis fascia will be used to close the perforation of ear drum. Gelfoam soaked in ciprofloxacin (0.3%) ear drops will be placed over the graft. Then ribbon gauze impregnated with Bismuth Iodoform Paraffin Paste (BIPP) was packed in external auditory canal above gelfoam. Skin incisions will be sutured in layers with 4-0 Vicryl and skin with 4-0 Ethilon. Mastoid bandage will be then applied.

After surgery patient will be shifted to ward, analgesics will be given routinely and on demand of the patient. First dressing will be done on first postoperative day, second dressing will be done on 3rd postoperative day and 3rd dressing on 6th postoperative days. Suture will be removed on sixth postoperative day and ear pack will be removed on tenth postoperative day. Any complication will be noted. Antibiotic ear drop Ciprofloxacin 3 drops 8 hourly will be prescribed for 2 weeks after the removal of pack. Wound Examination will be done on 1st, 2nd and 4th week by examining pinna, incision site and ear canal for any signs of infections. Graft status was assessed at 3 months for successful graft uptake or residual perforation

Benefit of participation:

You will have the opportunity to be the first to benefit from a new method under study. You will have the chance to play an active role in your own health care and gain a greater understanding of your disease or condition. You will help society by contributing to medical research. Even if you don't directly benefit from the results of the clinical trial you take part in, the information gathered can help others and adds to scientific knowledge. People who take part in clinical trials are vital to the process of improving medical care. There are no reported side effects of the treatment methods.

Funding the study:

The funding of this study will be done by the researcher and the hospital where this study will be carried out.

Privacy:

Your name will not be published anywhere that data about the trial are published or included in any publicly available information.

ELIGIBILITY:
Inclusion Criteria:

* Age : patients between 6 to 15 years of age
* Gender : both male and female patients
* Disease: Chronic otitis media mucosal inactive (dry for at least 4 weeks)

Exclusion Criteria:

* Actively discharging ear pre-operatively
* Revision myringoplasty
* Allergic to co-amoxiclav

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2015-06-06 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
: Number of Participants with postoperative wound infection | At Visit 1, [Post-op Day 1 ], at Visit 2 [Post-op Day 3] ,at Visit 3 [Day 8 to Day 14] ], at Visit 4 [ Day 28 to day 30]
  Number of participants who have had at least one episode of infection in the postoperative period.
  postoperative infection : Infection occurring within 4 weeks of postoperative periods
  Postoperative infection : Presence of any of the following findings on clinical examination
  1. Wound gaping
  2. Purulent discharge from incision site
  3. Purulent discharge from external auditory canal
  Measurement tool used to assess the measure
  * Clinical examination of patient by examiner
  * Wound assessment : Examination of pinna , incision site and graft donor site
  * Any signs of infections if present will be noted in performa.

SECONDARY OUTCOMES:
Number of Participants with successful graft uptake | At Visit 4 [ Day 28 to day 30], at Visit 5 [ day 80 to day 90]
  Number of participants who have had successful graft uptake at the end of 3 months of postoperative period
  Successful graft uptake: complete healing of tympanic membrane and graft is intact.
  Graft uptake failure : perforation of any size Measurement tool used to assess the measure
  * otoscopic examination of the operated ear
  * Successful Graft uptake or failure is noted on performa.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Khanal, MS,ENT, Principal Investigator — Ganesh Man Singh Memorial Academy (GMSMA) of ENT-Head and Neck Studies, TU Teaching Hospital, Institute of Medicine (IOM)

REFERENCES:
- [Derived] Khanal P, Guragain RP, Bhusal CL. Comparison of postoperative infection and graft uptake rate using single dose of intravenous co-amoxiclav versus no antibiotic in children undergoing myringoplasty: A randomized controlled trial. Int J Pediatr Otorhinolaryngol. 2020 Apr;131:109893. doi: 10.1016/j.ijporl.2020.109893. Epub 2020 Jan 18. PMID 31981921